CLINICAL TRIAL: NCT02659111
Title: Effects of Physical Training in Shunt-operated Patients With Idiopathic Normal Pressure Hydrocephalus
Brief Title: Effects of Physical Training in iNPH
Acronym: iNPhys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Fredrik Lundin, MD, PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dnr 205/250-31
Record Dates: First submitted 2016-01-12; First posted 2016-01-20 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Hydrocephalus, Normal Pressure
Keywords: Exercise Therapy
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-intensity physical exercise, HIFE (Experimental)
  Interventions: Other: High Intensive Functional Exercise (HIFE); Other: Physical training advice
- Physical training advice (Active Comparator)
  Interventions: Other: Physical training advice

INTERVENTIONS:
Other: High Intensive Functional Exercise (HIFE) — Patients invited to high-intensity physical exercise, HIFE by a physiotherapist with special competence in neurology at one of the two centers, or by a general physiotherapist where the patient lives. Goal Attainment Scaling is performed. The training will be given twice a week for one hour during 12 weeks . At least 18 of 24 training session in a four month period of time will be required. A training manual will be distributed to each training physiotherapist. The patients will also be encouraged to do additional training and they will receive standardized written physical training advice
  Arms: High-intensity physical exercise, HIFE
Other: Physical training advice — Patients randomized to written advice for physical training will be given a leaflet with instructions how to train by there own.The physiotherapist responsible for evaluating sets goals together with the patient according to Goal Attainment Scaling.

SUMMARY:
Patients with idiopathic Normal Pressure Hydrocephalus (iNPH) have variable difficulties regarding gait, balance, cognition and micturition. A shunt operation will improve these difficulties in most cases. Data suggest however, that they do not change their physical activity postoperatively. Physical training has been shown to be beneficial in patients with similar diseases i.e. Parkinson. The aim of this study is to apply a high intensity physical training program after a shunt operation to see if the patients can improve their physical capacity and ambulatory activity more than patients who only receive standardized written advice about physical training.

DETAILED DESCRIPTION:
Consecutive patients with iNPH at the neurological departments of University Hospital of Linköping and at Sahlgrenska University Hospital are included and randomized for either physical training according to a validated training concept for elderly and cognitive impaired patients named HIFE ( High Intensity Functional Exercise) together with a standardized written instruction for home training of physical exercises or only a standardized written instruction for home training. Goal Attainment Scaling will be used to set measurable goals together with the patient. The training will take place in a facility where physiotherapists are available either at the two centers or close to the patient´s home.Those physiotherapists at the centers responsible for the training will contact and send the local physiotherapists a manual and give instructions about the HIFE concept and will also stay in contact for the whole intervention i.e. 12 weeks ( one hour two times a week). A minimum of 18 out of 24 session will be required.

ELIGIBILITY:
Inclusion Criteria:

Shunt-operated patients with Idiopathic Normal Pressure Hydrocephalus diagnosed according the international guidelines from 2005

Exclusion Criteria:

MMSE: equal to and below 16 and/or inability to walk, with or without support , for 10 m.

Other disease, e.g severe heart disease, asthma making intensive physical training impossible.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in iNPH-scale | 3 and 6 months postoperatively
  iNPH-scale (Hellström et al) is a validated scale consisting of four domains; balance, gait, cognition and micturition to evaluate severity of iNPH.
Change in GAS | 3 and 6 months postoperatively
  Goal Attainment Scaling. A goal i set and an assessment is made according to a five-graded scale defining in what degree the goal is achieved.

SECONDARY OUTCOMES:
Quality of life | 3 and 6 months postoperatively
  EQ-5D-5L
Depression | 3 and 6 months postoperatively
  Beck Depression Inventory II
Disability | 3 and 6 months postoperatively
  Modified Rankin Scale
Muscle strengths | 3 and 6 months postoperatively
  The test is called "Chair-stand test". Leg strengths is measured, by counting number of raising ups from sitting to standing, that the research person is able to in 30 sec.
Physical endurance test | 3 and 6 months postoperatively
  Testing the distance a person is able to walk in 6 min
Falls | 3 and 6 months postoperatively
  Registration of the actual number of falls in the last three months
Actigraphy | 3 and 6 months postoperatively
  Actigraphy is a method to evaluate physical activity in a research person´s normal life. SenseWear is used to record number of steps daily but also time spent lying and standing which will give information about the activity.
Balance | 3 and 6 months postoperatively
  Timed Up and Go
ADL | 3 and 6 months postoperatively
  ADL taxonomy
Activity | 3 and 6 months postoperatively
  Grimby 6
Life satisfaction | 3 and 6 months postoperatively
  LiSat 11 is a validated questionnaire with 11 items concerning different aspects of quality of life,.
Diurnal rhythm | 3 and 6 months postoperatively
  Actigraphy (SenseWear) is used for one week. Diurnal rhythm will be assessed by measuring the peak amplitude of acitivity daily, the mean amplitude of activity daily and the 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Lundin, MD, PhD, Principal Investigator — Dept of Neurology
Locations (1):
- Dept of Neurology, Linköping, Sweden

REFERENCES:
- [Derived] Rydja J, Kollen L, Ulander M, Tullberg M, Lundin F. Physical Capacity and Activity in Patients With Idiopathic Normal Pressure Hydrocephalus. Front Neurol. 2022 Mar 28;13:845976. doi: 10.3389/fneur.2022.845976. eCollection 2022. PMID 35418936
- [Derived] Rydja J, Kollen L, Hellstrom P, Owen K, Lundgren Nilsson A, Wikkelso C, Tullberg M, Lundin F. Physical exercise and goal attainment after shunt surgery in idiopathic normal pressure hydrocephalus: a randomised clinical trial. Fluids Barriers CNS. 2021 Nov 22;18(1):51. doi: 10.1186/s12987-021-00287-8. PMID 34809666